CLINICAL TRIAL: NCT05462509
Title: Feasibility of Use of the PATH bCPAP Kit Including Oxygen Blenders in a Neonatal Population in Uganda
Brief Title: Feasibility of Use of the PATH bCPAP and Oxygen Blenders Device With Neonates in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: University of Washington (Other); Adara Development (Unknown); Kiwoko Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1519912-11
Record Dates: First submitted 2022-06-16; First posted 2022-07-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Distress Syndrome; Infant, Premature
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bCPAP and blenders (Experimental): all patients admitted to the newborn care unit with respiratory failure will be evaluated for treatment with bCPAP per unit standards. All patients that meet treatment criteria will receive bCPAP. Patients for whom consent is available will be enrolled and start bCPAP therapy with the PATH kit. Patients for whom consent is not given or not available will start Kiwoko bCPAP. Patients who began bCPAP therapy with the Kiwoko kit and obtain consent within 24 hours of starting their bCPAP therapy may switch from Kiwoko to PATH bCPAP. Patients with >24 hours of Kiwoko bCPAP therapy are no longer eligible for enrolment. , oxygen blending for patients treated with PATH bCPAP will occur by the following two methods- and will be used in this order of preference:
  1. blending via air compressor (standard of care in unit and used when available)
  2. blending via PATH blender (when no compressor available)
  Interventions: Device: bCPAP with blenders

INTERVENTIONS:
Device: bCPAP with blenders — The intervention device is a low-cost bCPAP kit which includes two fixed-ratio oxygen blenders that do not require a source of pressurized air. These simple and inexpensive devices sit in-line from the oxygen source and dilute the flowing stream of oxygen with room air, obviating the need for a pressurized source of air. The oxygen may be supplied from either high-pressure sources or low-pressure sources such as oxygen concentrators. Each of the two blenders are single plastic parts, injection moulded from a biocompatible, medical-grade polyethylene resin. No electricity is required for the blenders to provide a stable and constant mix of air and oxygen over the full range of clinically relevant pressure and flows for newborns.

SUMMARY:
In this mixed methods study, the investigators assessed feasibility of use of the PATH bCPAP kit on neonatal patients as well as the usability and acceptability of the device by healthcare workers.The study took place in a rural Ugandan special care nursery with experience in bCPAP. Neonates with respiratory failure were consented and treated with the PATH bCPAP kit and blenders. The investigators conducted prospective data collection of the device use through observation as well as collected qualitative data via interviews with nurses, which were analyzed using a rapid qualitative analytical method.

DETAILED DESCRIPTION:
Preterm birth is responsible for 1/3 of deaths under age five- the majority which occur in resource-constrained settings. Many of these deaths are due to respiratory failure which can be treated with bubble continuous positive airway pressure (bCPAP). Commercialized bCPAP devices are expensive, leading resource-constrained settings to make and use improvised devices. These improvised devices have not been tested for performance and run on 100% oxygen. WHO guidelines strongly advise against the use of 100% oxygen-particularly with preterm newborns where it can cause blindness, lung and brain injury.

To address this need, PATH has developed a low-cost bCPAP kit which includes oxygen blenders that do not require electricity nor a source of pressurized air to blend oxygen with air. The objectives of this early feasibility study are to:

1. assess the operational feasibility of using the PATH bCPAP kit including, when appropriate, in-line oxygen blending on neonatal patients and
2. assess the usability and acceptability of the PATH bCPAP kit with oxygen blenders by healthcare workers.

Newborns will be treated with the PATH bCPAP kit and a subset of these will also be treated with the PATH blender as needed to provide blended oxygen. Results from this study will be used to identify appropriate modification to the use procedures and/or the device as needed. Once testing is completed and product revision finalized, the PATH kit and blenders will allow resource-constrained settings to provide rigorously tested bCPAP therapy and blended oxygen to patients with reduced risk of morbidity from oxygen toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Newborns <44 weeks post menstrual age with respiratory failure requiring treatment with bCPAP therapy during the period of study
* Parent or legal guardian consented to participation in the study within 24 hours of bCPAP initiation.

Exclusion criteria:

* No parental nor legal guardian consent for participation in the study.

Ages: 24 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Usability of the bCPAP device | Immediately after use of the device
  Median time of device set up in minutes
Usability of the blenders device | Immediately after use of the device
  Median time of changing blender in seconds
Acceptability of the bCPAP and blenders device | Within the first five days of having used the device for the first time
  Median score on Likert-type scale (rating of 1-10 with 10 being best) for health worker satisfaction with device

SECONDARY OUTCOMES:
Demographics of patients treated | At enrollment
  Place of birth, sex, median weeks gestation
Clinical characteristics of patients treated: median admission weight | At enrollment
  Median admission weight in kg
Clinical characteristics of patients treated: reason for admission | At enrollment
  Reason for admission
Outcomes of patients treated: patient age | At baseline
  Age (in weeks) when bCPAP therapy started
Outcomes of patients treated: device pressure | Immediately at end of bCPAP therapy
  Median pressure (in cmH2O) used during treatment
Outcomes of patients treated: device flow | Immediately at end of bCPAP therapy
  Median oxygen source flow (in LPM) used during treatment
Outcomes of patients treated: treatment length | Immediately at end of bCPAP therapy
  Median treatment length in days

CONTACTS AND LOCATIONS:
Locations (1):
- Kiwoko Hospital, Kiwoko, Nakaseke, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hedstrom AB, Nyonyintono J, Saxon EA, Nakamura H, Namakula H, Niyonshaba B, Nakakande J, Simpson N, Vaughan M, Wollen A, Mubiri P, Waiswa P, Coffey PS, Batra M. Feasibility and usability of a very low-cost bubble continuous positive airway pressure device including oxygen blenders in a Ugandan level two newborn unit. PLOS Glob Public Health. 2023 Mar 8;3(3):e0001354. doi: 10.1371/journal.pgph.0001354. eCollection 2023. PMID 36963078

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT05462509/Prot_SAP_000.pdf